CLINICAL TRIAL: NCT03111836
Title: Effectiveness of User and Expert Driven Internet-based Lifestyle Interventions on Hypertension Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, sam liu, Researcher, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UT01
Record Dates: First submitted 2017-04-04; First posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Sham Comparator): The Control group received limited to general information on blood pressure management
  Interventions: Behavioral: Control Group
- Expert-driven group (Active Comparator): The intervention will consisted of pre-determined exercise and dietary goals (e.g. increase daily steps by 1000 steps, consuming 2-3 servings of fruit and vegetables per day).
  Interventions: Behavioral: Expert-Driven Group
- User-driven group (Active Comparator): The User-driven group received an intervention that enabled participants to select their areas of lifestyle change using text and video web links embedded in the email. The trans-theoretical model was used to inform the design of the User-driven program.
  Interventions: Behavioral: User-driven group

INTERVENTIONS:
Behavioral: Control Group — Received general information about blood pressure control. All subjects will be sent 16 e-messages on a weekly schedule.
  Arms: Control group
Behavioral: Expert-Driven Group — The user-driven e-Counselling group will receive a lifestyle program where the user are able to choose areas of focus. All subjects will be sent 16 e-messages on a weekly schedule.
  Arms: Expert-driven group
Behavioral: User-driven group — The user-driven e-Counselling group will receive a lifestyle program where the user are able to choose areas of focus. All subjects will be sent 16 e-messages on a weekly schedule.
  Arms: User-driven group

SUMMARY:
Hypertension is a leading risk factor for cardiovascular disease and mortality. Lifestyle counseling is recommended as a first line therapy for reducing blood pressure (BP) and risk for cardiovascular events. Recent studies suggest that e-based lifestyle interventions are effective in evoking therapeutic change in BP1. However, BP response and adherence to exercise and diet behavior varies significantly after e-based interventions due to variations in treatment methodologies. Consensus is not yet established for a standardized e-counseling protocol for hypertension. As noted in our systematic review, the two dominant models of e-counseling procedures are expert-driven (protocol driven, prescriptive) and user-driven (self-guided, collaborative). Expert-driven programs prescribe specific changes for lifestyle behavior which are intended to facilitate compliance to behavioral change. In contrast, the user-driven method actively involves the subject in goal-setting and/or the selection of the intervention used to reach the behavioral goal. One conclusion from the systematic review is that these models are used indiscriminately in e-counseling programs. There is currently inadequate data to determine the efficacy of programs that are expert-driven vs. user-driven in reducing BP while modifying lifestyle behaviour. It is possible that a combination of expert-driven and user-driven features for lifestyle e-counseling is most effective. However, before these two approaches can be combined, it is essential to establish the strengths and limitations of each model.

DETAILED DESCRIPTION:
This study will use a 3-parallel group, randomized controlled design: 3 (Groups: Control, expert-driven, and user-driven e-Counselling) by 2 (Assessments: baseline, 4-month). Controls will receive general e-information on BP management. The expert-driven e-Counselling group will provide a prescribed exercise and a diet plan. The user-driven e-Counselling group will a program that enables the patient to choose areas of focus. All subjects will be sent 16 e-messages on a weekly schedule.

ELIGIBILITY:
Inclusion Criteria:

* Unchanged prescription for anti-hypertensive medication at least 2 months before enrollment.
* Participants prescribed antihypertensive medication were also required to have SBP ≥130 mmHg and/or DBP ≥85 mmHg, in order to prevent "floor effects".

Exclusion criteria included:

* Diagnosis of kidney disease, major psychiatric illness (e.g. psychosis), alcohol or drug dependence in the previous year, pregnancy and sleep apnea. There was no racial or gender bias in the selection of participants.

Ages: 35 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2014-07-01 (Actual); Study Completion 2015-06-01 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure | Change from Baseline Systolic Blood Pressure at 4 months

SECONDARY OUTCOMES:
Diastolic Blood Pressure | Change from Baseline Diastolic Blood Pressure at 4 months
Blood Lipids (HDL, LDL, Cholesterol) | Change from Baseline Blood Lipids (HDL, LDL, Cholesterol) at 4 months
Fruit and Vegetables | Change from Baseline Daily servings of Fruit and Vegetables at 4 months
  Diet History Questionaire
Daily Steps | Change from Baseline Daily Steps at 4 months
  Pedometer

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu S, Brooks D, Thomas SG, Eysenbach G, Nolan RP. Effectiveness of User- and Expert-Driven Web-based Hypertension Programs: an RCT. Am J Prev Med. 2018 Apr;54(4):576-583. doi: 10.1016/j.amepre.2018.01.009. Epub 2018 Feb 16. PMID 29456025